CLINICAL TRIAL: NCT02918422
Title: Controlled Feeding Study to Show Effects of Manipulating Carbohydrate and Cheese on Health Markers In Individuals With Metabolic Syndrome
Brief Title: Controlled Clinical Study to Determine Novel Health Benefits of Cheese Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jeff Volek, Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GRT00036921; 60047084 (Other Grant/Funding Number: Dairy Management Inc)
Record Dates: First submitted 2016-02-25; First posted 2016-09-29 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Metabolic Syndrome X
Keywords: Diet Intervention; Metabolic Syndrome; Feeding Study; Prediabetes
MeSH Terms: conditions — Metabolic Syndrome; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- High Carbohydrate No Cheese (Experimental): Intervention: Nutritional and Dietary Manipulation. This arm will be provided food with an approximate macronutrient breakdown of: 55% CHO, 20% PRO and 25% fat with ~6oz Cheese (gouda or cheddar) per day being used as a fat source.
  Interventions: Other: Nutritional and Dietary Manipulation
- High Carbohydrate High Cheese (Experimental): Intervention: Nutritional and Dietary Manipulation. This arm will be provided food with an approximate macronutrient breakdown of: 55% CHO, 20% PRO 25% and Fat 25% with ~6oz Cheese (gouda or cheddar) per day being used as a fat source.
  Interventions: Other: Nutritional and Dietary Manipulation
- Mod. Carbohydrate High Cheese (Experimental): Intervention: Nutritional and Dietary Manipulation. This arm will be provided food with an approximate macronutrient breakdown of: 30% CHO, 20% PRO and 50% Fat with ~6oz Cheese (gouda or cheddar) per day being used as a fat source.
  Interventions: Other: Nutritional and Dietary Manipulation
- Low Carbohydrate High Cheese (Experimental): Intervention: Nutritional and Dietary Manipulation. This arm will be provided food with an approximate macronutrient breakdown of: 10% CHO, 20% PRO and 70% Fat with ~6oz Cheese (gouda or cheddar) per day being used as a fat source.
  Interventions: Other: Nutritional and Dietary Manipulation

INTERVENTIONS:
Other: Nutritional and Dietary Manipulation — Participants will undertake a controlled feeding intervention. All food will be prepared and delivered to participants by research staff. Participants will be asked to exclusively eat what is provided to them in efforts to control any dietary effects.

SUMMARY:
To determine the effects of high cheese diets varying in carbohydrate content on markers of disease risk.

DETAILED DESCRIPTION:
Summary of Proposed Research:

This project will involve four controlled 4 wk feeding periods in individuals with metabolic syndrome (currently 1/3 of US adults). After a 2 wk run-in period, 20 subjects will be fed one of three diets in a randomized and balanced order: a typical American High-Carb diet high in cheese (6 oz/day), a High-Carb diet low in cheese (0 oz/day), or a Moderate-Carb, high-cheese diet (6 oz/day), Low-Carb, high cheese where cheese displaces an isocaloric amount of carbohydrate. There will be a 2 wk washout period separating trials during which subjects consume their normal diet. Specific menus will be designed for each feeding phase and all food will be prepared for subjects. Testing will occur at baseline and after each feeding period. Measures of cholesterol beyond standard LDL- and HDL-cholesterol will be done by examining lipoprotein particle size, apolipoproteins, and fatty acid composition [i.e., accumulation of saturated fat in blood and tissues, palmitoleic acid (highly linked to cardiovascular disease), and detection of phytanic acid (a uniquely bioactive fatty acid in dairy fat)]. Changes in whole body and regional fat, including measures of visceral fat and liver fat, will be examined non-invasively by dual-energy X-ray absorptiometry (DXA) and magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference (≥101.6 cm men, ≥88.9 cm women)
* Blood pressure (≥130/85 mm Hg) or current use of antihypertensive medication
* Fasting plasma glucose (≥100 mg/dL)
* Triglycerides (≥150 mg/dL)
* HDL-C (<40 mg/dL men, <50 mg/dL women)

Exclusion Criteria:

* Hypercholesterolemia
* Diabetes
* Liver, kidney or other metabolic or endocrine dysfunction, gastrointestinal disorders
* Regular smokers
* Lactose-intolerant
* Consume excessive amounts of alcohol (>3 drinks/d)
* Have used cholesterol, diabetic, antibiotic or antifungal medications in the past 3 months
* Women who are pregnant or lactating
* Participants taking any probiotics or supplements known to affect serum lipid levels, inflammation, antioxidant status or the gut microbiota will be asked to discontinue use to allow for washout of any metabolic effects.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09; Primary Completion 2018-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Plasma Fatty Acid Composition and Lipoprotein Analysis | Through study completion, an average of 2 years.
  Blood analysis for Fatty Acid Composition and Lipoproteins will by conducted by Lipid Technologies and Quest Diagnostics, respectively.

SECONDARY OUTCOMES:
Change in Body Composition as Assessed by DEXA and MRI | Through study completion, an average of 2 years.
  Participants will undergo both DEXA and MRI scans, conducted by trained professionals. DEXA will be used to determined subcutaneous adiposity. MRI post-imaging analyses will determine both hepatic and visceral fat content.
Change in Blood-based Inflammation Markers | Through study completion, an average of 2 years.
  Inflammatory biomarkers in the blood will be assessed using a Multiplex ELISA system. The inflammatory markers to be measured are: IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12, IL-13 and TNF-α.
Change in Blood Metabolite Profiles | Through study completion, an average of 2 years.
  NMR spectroscopy (600 Mhz) will be used to obtain metabolic profiles of serum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Volek, PhD, Principal Investigator — Ohio State University
Locations (1):
- Physical Activity and Education Services - PAES, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Final results will be published via peer-review process.

REFERENCES:
- [Derived] Hyde PN, Sapper TN, Crabtree CD, LaFountain RA, Bowling ML, Buga A, Fell B, McSwiney FT, Dickerson RM, Miller VJ, Scandling D, Simonetti OP, Phinney SD, Kraemer WJ, King SA, Krauss RM, Volek JS. Dietary carbohydrate restriction improves metabolic syndrome independent of weight loss. JCI Insight. 2019 Jun 20;4(12):e128308. doi: 10.1172/jci.insight.128308. eCollection 2019 Jun 20. PMID 31217353